CLINICAL TRIAL: NCT06169904
Title: B7-Family Score Predicts Clinical Outcome From Chemotherapy and Checkpoint Blockade for Patients With Urothelial Carcinoma
Brief Title: B7-Family Score in Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fudan University (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: FUDAN-BLCA-01
Record Dates: First submitted 2023-11-29; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Cisplatin; atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed, paraffin embedded samples have been constructed into TMA to evaluate protein expression within the tissue.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cisplatin injection — We observed the UC patients from Zhongshan Hospital receiving or not receiving adjuvant cisplatin-based chemotherapy after radical cystectomy.
  Other Names: Atezolizumab injection

SUMMARY:
Immunotherapy has been found to confer substantial survival benefits to the patients with higher mutation burdens, which become the first biomarker approved by FDA in urothelial carcinoma (UC). Nevertheless, among the patients with high mutation burdens, some still remained refractory to immunotherapy. The B7 family molecules have long been perceived as vital determinant of immune response and may define dominant molecular subsets associated with immunotherapeutic response. Simultaneously, our previous study (Eur J Cancer. 2022,171:133-142) unveiled the potential of B7-H4 as a candidate biomarker to refine the predictive capability of tumor mutation burden (TMB) in immunotherapeutic efficacy based on its significant correlation with TMB in MIBC. We hypothesized that the integration of B7 family molecules with TMB could better identify patients with better response to checkpoint blockade.

In this retrospective study, a total of 1,084 UC patients from 5 independent cohorts were enrolled. We established the B7 Family Score (BFS) by the expression patterns of three B7 family members: PD-L1 (CD274), B7-H3 (CD276) and B7-H4 (VTCN1) based on protein and transcriptomic level respectively. We further investigated the correlation of BFS with genomic features and therapeutic response in UC. In addition, we integrated the BFS with tumor mutation burden (TMB) to better stratify the clinical benefit from PD-L1 blockade and platinum-based chemotherapy.

DETAILED DESCRIPTION:
On the basis of established findings in the prognostic and functional properties of the three B7 family members, i.e., PD-L1, B7-H3, and B7-H4, we employed the IMVigor210 cohort as the discovery cohort to establish the concept of B7 Family Score (BFS). To maximize the prognostic value of the system, we introduced the R package survMisc (0.5.5) in the IMvigor210 cohort to determine the best cut-off value of mRNA expression level of the B7 family members (i.e. CD274, CD276, and VTCN1) by calculating the minimum log-rank P value accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with muscle-invasive bladder cancer receiving radical cystectomy have been included in this study.

Exclusion Criteria:

* Patients with non-muscle invasive bladder cancer were not eligible in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Among the 215 patients originally diagnosed with bladder cancer who underwent radical cystectomy at Zhongshan Hospital of Fudan University from 2002 to 2014, eighty-seven patients were excluded: 60 patients without muscle-invasive bladder cancer (MIBC), 13 patients with non-urothelial carcinoma, and 36 specimens with dots lost on the tissue microarray (TMA) during the immunohistochemistry (IHC) assay. Therefore, 106 patients are enrolled in the ZSHS cohort, 51 of whom received adjuvant cisplatin-based chemotherapy which lasted at least one therapeutic cycle. The overall survival (OS) and the recurrence-free survival (RFS) were defined as the period from the date of RC to the date of death or first recurrence, or to the latest follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Death | 1/1/2002-1/1/2022
  The time when patients died is the primary outcome measure.